CLINICAL TRIAL: NCT00814827
Title: Mycobacterial and Opportunistic Infections in HIV-Negative Patients Associated With Autoantibodies to Interferon-gamma
Brief Title: Mycobacterial and Opportunistic Infections in HIV-Negative Thai and Taiwanese Patients Associated With Autoantibodies to Interferon-gamma
Status: Active, not recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999909060; 09-I-N060
Record Dates: First submitted 2008-12-24; First posted 2008-12-25 (Estimated); Last update posted 2025-12-23 (Actual); Status verified 2025-07-08

CONDITIONS: Nontuberculous Mycobacteria; Mycobacterium Tuberculosis; Opportunistic Infections
Keywords: Interferon-Gamma; Autoantibodies; Disseminated Infection; Pulmonary Infection; Blood Donor; Natural History
MeSH Terms: conditions — Opportunistic Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Group 1: Patients with nontuberculous mycobacteria (NTM) alone.
- Group 2: Patients with non-NTM opportunistic infection, either with or without concurrent NTM infection.
- Group 3: Patients with pulmonary mycobacterium tuberculosis (MTB).
- Group 4: Patients with disseminated mycobacterium tuberculosis (MTB).
- Group 5: Blood Specimen Donors.

SUMMARY:
Opportunistic infections are caused by bacteria, mycobacteria, fungi or viruses that do not normally cause infections in people with healthy immune systems. Some of these infections can cause public health concerns, especially in areas with limited access to treatment. People who acquire opportunistic infections usually have diseases that affect their immune systems, such as human immunodeficiency virus (HIV), or do not have enough white blood cells to fight the infection. However, some people acquire opportunistic infections even though they have normal amounts of white blood cells and are free from known diseases that harm their immune systems. This study will investigate some of the reasons that otherwise healthy people get opportunistic infections to learn more about why some people are more likely to have them.

This study will include up to 210 HIV-negative males and females older than 18 years of age who have opportunistic infections. The patients will be drawn from multiple sites in Thailand and Taiwan including Khon Kaen University Hospital, Siriraj Hospital, Ramathibodi Hospital, National Taiwan University Hospital, National Cheng-Kung University Hospital

Patients will undergo an initial evaluation that will include a physical examination, medical history, and blood and urine testing. Additional tests will be conducted if the researchers consider that the tests are medically necessary to treat the opportunistic infection; the results of the tests will be reviewed and saved for study purposes. Depending on the severity of the infection, the initial evaluation may take more than 1 day to complete.

After the evaluation, patients will be given standard and appropriate medicines to treat the infections.

Patients will return for follow-up visits to allow researchers to monitor their condition and to assess how well the patient is responding to the treatment. Patients will be evaluated by the study researchers at least once a year for 2 years following the initial treatment.

DETAILED DESCRIPTION:
The acquisition of opportunistic infections has been causally linked to innate and acquired immunodeficiencies. We have recently identified a population of Asian women with autoantibodies to interferon gamma (IFN?), all of whom were diagnosed by virtue of nontuberculous mycobacterial infections. Similar patient populations have been reported from Thailand, and we have found similar autoantibodies in anonymous serum samples from there. In addition, many of the Thai patients who have disseminated or lymphatic nontuberculous infections have had other opportunistic infections (OI), such as salmonella, penicilliosis, and histoplasmosis. However, they have normal lymphocyte counts and are human immunodeficiency virus (HIV) negative. Therefore, the identification of autoantibodies to a critical cytokine, the occurrence of opportunistic infections, and the lack of other common explanations suggests that this is an important population to study. We propose to enroll patients in a natural history study of non-HIV opportunistic infections to explore the presence of autoantibodies to cytokines, and to examine potential immunogenetic factors influencing the development of this disease. Plasma, cells, and DNA samples will be obtained and stored for use in this study. This study will accrue up to 265 patients over 5 years as per the protocol with follow up for 15 years on each patient, sample size justification and the groups described in the protocol.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients must meet all of the following criteria at the time of evaluation to be eligible for enrollment into the study cohorts:

Group 1 (NTM alone):

1. Past or current infection with NTM proven by culture or specific DNA detection in the presence of a compatible clinical picture as judged by the responsible clinician and PI on site.
2. NTM is not felt to iatrogenic (such as indwelling catheter associated or post-operative wound infection)
3. HIV negative within 3 months either prior to the diagnosis of OI, or prior to enrollment in this study, if HIV status was unknown at the time of OI
4. No evidence of active malignancy
5. No systemic corticosteroids at time of diagnosis of OI (defined as greater than 4 weeks at a dose greater than 10 mg per day of prednisone within 3 months prior to diagnosis of the NTM)
6. No preexisting immune deficiency

Group 2 (non-NTM OI with or without NTM):

1. Patients must have or have had proven infection with one or more of the following organisms: disseminated Salmonella, Listeria, Penicillium, Burkholderia pseudomallei, Cryptococcus, Histoplasma, Herpes zoster involving 2 or more non-contiguous dermatomes, or extradermal involvement or other opportunistic infections not listed above, but relevant, as determined by the PI.
2. Patient may have infection with NTM in addition to one or more of the above infection(s).
3. HIV-negative within 3 months either prior to the diagnosis of OI, or prior to enrollment in this study, if HIV status was unknown at the time of OI diagnosis
4. No evidence of active malignancy
5. No systemic corticosteroids at time of diagnosis of OI (defined as greater than 4 weeks at a dose greater than 10 mg per day of prednisone within 3 months prior to diagnosis of the NTM)
6. No preexisting immune deficiency

Group 3 (diseased control with pulmonary MTB):

1. Active pulmonary MTB, i.e. patients who have sputum that is either culture positive for MTB or AFB positive and responding to therapy for MTB.
2. Diagnosed with the past 6 months.
3. No concurrent infections due to NTM or OI listed under above inclusion criteria for study subjects
4. No clinical evidence of HIV

Group 4 (diseased control with disseminated MTB):

Disseminated MTB includes infections involving greater than or equal to 2 noncontiguous sites, one of which may include pulmonary disease or greater than or equal to 2 separate groups of lymph nodes.

1. Active disseminated MTB or cured disseminated MTB
2. No concurrent infections due to NTM or OI listed under above inclusion criteria for study subjects
3. HIV negative within 3 months either prior to the diagnosis of MTB, or prior to enrollment in this study, if HIV status was unknown at the time of MTB diagnosis
4. No evidence of active malignancy
5. No systemic corticosteroids at time of diagnosis of OI (defined as > 4 weeks at a dose > 10 mg per day of prednisone within 3 months prior to diagnosis of the NTM)
6. No preexisting immune deficiency.

Group 5 (Blood Specimen Donors):

Eligibility criteria not applicable. Blood will be collected from volunteers, and no medical evaluation will be performed.

To be a blood donor the person cannot be excluded per the exclusionary criteria:

1. Patient < 18 or > 85
2. Weight > 45 kg (99 lbs)
3. Receiving chemotherapy of have cancer
4. Receiving immunosuppressant medications
5. Have a history of heart, lung, kidney disease of bleeding disorder.

EXCLUSION CRITERIA:

Patients will be excluded for the following reasons:

1. HIV-positive serostatus for groups 1, 2 and 4 (groups 3 and 5 will not be routinely performing HIV testing)
2. Active malignancy
3. Medical conditions requiring immune modulating therapy (i.e. corticosteroids, biological agents, anti-metabolites) and /or chemotherapy
4. Any other medical conditions unsuitable for this study as determined by the principal investigator
5. Age less than 18 years
6. Receiving any other investigational study agents when enrolling on this study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective natural history cohort study with a case-control component. Patients will be recruited from 5 groups: 1) subjects with NTM alone, 2) subjects with a non-NTM OI, either with or without concurrent NTM infection, 3) subjects with pulmonary MTB, 4) subjects with disseminated MTB, and 5) Blood Specimen Donor controls.
Sampling Method: Non-Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2010-01-07 (Actual)

PRIMARY OUTCOMES:
Identification of the presence of autoantibodies to IFNy in HIV-negative Thai and Taiwanese patients with disseminated NTM and OI who are followed at the participating institutions. | ongoing
  Compare the baseline prevalence rate of autoantibodies to IFNg, as defined by having >75% inhibition, in patients with disseminated NTM or other OI (groups 1 and 2) versus normal or diseased controls (groups 3 and 5).

SECONDARY OUTCOMES:
Identification of predisposing factors for the development of autoimmunity to cytokines and/or their receptors. | ongoing
  Identification of predisposing factors for the development of autoimmunity to cytokines and/or their receptors.
Identification of other autoantibodies that might manifest similarly to patients with autoantibodies to IFNg. | ongoing
  Identification of other autoantibodies.
Characterization of the natural history and specific microbiology in HIV-negative patients with disseminated NTM and other OI and to determine any statistically significant differences from MTB controls or healthy blood bank donors. | ongoing
  Characterization of the natural history and infections of consecutive patients with NTM alone and NTM with other OI. Speciation of the opportunistic infections identified and categorization of these infections with descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Christa S Zerbe, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (5):
- National Taiwan University, Taiwan, China
- National Cheng Kung University, Tainan, Taiwan
- Thailand (3):
  - National Siriraj Hospital, Mahidol Universtiy, Bangkok
  - Ramathibodi Hospital, Mahidol Universtiy, Bangkok
  - Srinagarind Hospital, Khon Kaen

IPD SHARING:
Plan to Share IPD: Yes
We will share human data generated in this study for future research as follows:@@@@@@@@@@@@ (Summation)Identified data in the Biomedical Translational Research Information System (BTRIS, automatic for activities in the NIH CC).@@@@@@@@@@@@ (Summation)De-identified or identified data with approved outside collaborators under appropriate agreements.@@@@@@@@@@@@ (Summation)Data sharing may be complicated or limited in certain cases by contractual obligations or agreements with outside collaborators, such as cooperative research and development agreements, clinical trial agreements, other restraints, etc.
Supporting Information: SAP
Time Frame: IPD and supporting information will be available after completion of the study.
Access Criteria: Data will be shared through:@@@@@@@@@@@@ (Summation)BTRIS (automatic for activities in the NIH CC).@@@@@@@@@@@@ (Summation)Approved outside collaborators under appropriate individual agreements.@@@@@@@@@@@@ (Summation)Publication and/or public presentations.@@@@@@@@@@@@Data might be shared before publication.@@@@@@@@@@@@The PI will review all requests for sharing data.

REFERENCES:
- [Background] Dorman SE, Holland SM. Interferon-gamma and interleukin-12 pathway defects and human disease. Cytokine Growth Factor Rev. 2000 Dec;11(4):321-33. doi: 10.1016/s1359-6101(00)00010-1. PMID 10959079
- [Background] Patel SY, Ding L, Brown MR, Lantz L, Gay T, Cohen S, Martyak LA, Kubak B, Holland SM. Anti-IFN-gamma autoantibodies in disseminated nontuberculous mycobacterial infections. J Immunol. 2005 Oct 1;175(7):4769-76. doi: 10.4049/jimmunol.175.7.4769. PMID 16177125
- [Background] Kampmann B, Hemingway C, Stephens A, Davidson R, Goodsall A, Anderson S, Nicol M, Scholvinck E, Relman D, Waddell S, Langford P, Sheehan B, Semple L, Wilkinson KA, Wilkinson RJ, Ress S, Hibberd M, Levin M. Acquired predisposition to mycobacterial disease due to autoantibodies to IFN-gamma. J Clin Invest. 2005 Sep;115(9):2480-8. doi: 10.1172/JCI19316. Epub 2005 Aug 25. PMID 16127458
- [Derived] Browne SK, Burbelo PD, Chetchotisakd P, Suputtamongkol Y, Kiertiburanakul S, Shaw PA, Kirk JL, Jutivorakool K, Zaman R, Ding L, Hsu AP, Patel SY, Olivier KN, Lulitanond V, Mootsikapun P, Anunnatsiri S, Angkasekwinai N, Sathapatayavongs B, Hsueh PR, Shieh CC, Brown MR, Thongnoppakhun W, Claypool R, Sampaio EP, Thepthai C, Waywa D, Dacombe C, Reizes Y, Zelazny AM, Saleeb P, Rosen LB, Mo A, Iadarola M, Holland SM. Adult-onset immunodeficiency in Thailand and Taiwan. N Engl J Med. 2012 Aug 23;367(8):725-34. doi: 10.1056/NEJMoa1111160. PMID 22913682